CLINICAL TRIAL: NCT04105855
Title: Cross-Sectional Survey of Plasmodium and Other Parasites in Pregnant Women and Infants Around Maferinyah, Guinea
Brief Title: Malaria Prevalence Around Maferinyah, Guinea
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999919141; 19-I-N141
Record Dates: First submitted 2019-09-25; First posted 2019-09-26 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Malaria
Keywords: Organism; Seasonal; Blood Smear; Burden; Infections; Natural History
MeSH Terms: conditions — Malaria; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Finger prick/heel stick samples and peripheral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Older Infants: Infants age 6-12 months presenting for routine healthy visits
- Pregnant Women: Women 18 years and older (and emancipated minors) presenting for routine antenatal visits

SUMMARY:
Background:

Many women in Sub-Saharan Africa get malaria while they are pregnant. Plasmodium falciparum is a parasite that can cause malaria. Placental malaria (PM) caused by P. falciparum can cause anemia or death in first-time mothers. In infants, it can cause low birth weight, premature birth, or other problems. Some women don t show any signs of having PM. This makes it harder to know if they might have it. Researchers want to learn how much the seasons affect the number of women and infants who get PM as well as the severity of the disease. To do this, they are going to test women and babies who visit a health center in Guinea.

Objective:

To learn the seasonal burden of P. falciparum infection in pregnant women and otherwise healthy infants.

Eligibility:

Pregnant women ages 18 years and older (or emancipated minors) and infants ages 6-12 months.

Design:

Participants will include women and infants who visit the health center in Maf(SqrRoot)(Registered Trademark)rinyah, Guinea, for routine care. They can take part only once per pregnancy.

For screening, mothers will talk about their medical history. They will talk about their past pregnancies and their current pregnancy. They will answer questions about where they live and what they do to keep from getting malaria. Babies will be screened with their medical history and demographic information.

Participants will also give a blood sample. Adults will have a finger stick. Children will have a heel stick. Or they will have blood taken from a vein.

Participation will last for 1 visit to the health center.

DETAILED DESCRIPTION:
Malaria caused by Plasmodium falciparum continues to be a global problem with devastating consequences, in particular for at-risk populations such as pregnant women and young infants. Pregnancy malaria is associated with low birth weight (LBW), maternal anemia, and gestational hypertension; both inflammation and the fetal response to infection may contribute to these poor outcomes. Placental malaria (PM) is caused by P. falciparum-infected erythrocytes that bind to the placental receptor chondroitin sulfate A (CSA) and sequester in the placenta, where they cause disease and may lead to death for the mother and her offspring. Women become resistant to PM as they acquire antibodies that target surface proteins of placental parasites. In areas of stable transmission, acute severe malaria syndromes are limited to children under 5 years of age. The pathogenesis of severe malaria remains poorly understood, although some evidence suggests that parasites causing severe malaria may express distinct antigens on the surface of infected erythrocytes. Thus, vaccines to prevent malarial disease may need to target distinct antigens in order to protect pregnant women or young children.

The primary hypothesis in this study is that the burden of P. falciparum infection around Maferinyah, Guinea is sufficient to support future studies of malaria pathogenesis and immunity. We plan to enroll 1050 pregnant women and 1050 infants into a cross sectional study that will be conducted in Maferinyah and neighboring areas, Guinea. Women presenting for routine antenatal visits and older infants presenting for routine healthy visits (e.g, vaccinations, vitamins) at the health center in Maf(SqrRoot)(Registered Trademark)rinyah will be offered enrollment. Samples collected from the women and infants will be examined for evidence of infection by Pla smodium and other parasitic diseases in order to assess prevalence in these important reservoir populations. For our primary outcome, we will determine the prevalence of P. falciparum infection in these two key demographic groups, including their annual and seasonal variations, as these data will form the basis to design future natural history or interventional studies at this site. For our secondary outcomes, we will determine the prevalence of other parasitic infections based on multiplexed serologic assessments of blood samples.

ELIGIBILITY:
* INCLUSION CRITERIA:

For pregnant women, a study participant must satisfy the following criteria to be enrolled in this study:

* Pregnant women greater than or equal to 18 years of age (or emancipated minors) reporting for routine antenatal care at the health center without acute illness
* The study participant understands the study and gives informed consent for participation
* Willingness to share a positive test result for malaria or helminths with the health center in Maf(SqrRoot)(Registered Trademark)rinyah so treatment can be initiated if necessary
* Willingness to allow stored laboratory specimens to be used for future research

For children, a study participant must satisfy the following criteria to be enrolled in this study:

* Children 6-12 months of age at time of visit presenting for routine care at the health center without acute illness
* The parent or guardian understands the study and gives informed consent for participation of their child
* Willingness of parent/guardian to share a positive test result for malaria or helminths with the health center in Maferinyah so treatment can be initiated if necessary
* Willingness of parent/guardian to allow stored laboratory specimens to be used for future research

EXCLUSION CRITERIA:

-Conditions that in the judgment of the Principal Investigator or Clinical Investigators could adversely impact the safety of the study participant, including conditions that may impair the ability of the participant or participant s parent/guardian to understand the study. All such exclusions and the reason for exclusion will be documented.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women 18 years of age and older (including emancipated minors) and 6-12 month old infants presenting for routine visits at Maf(SqrRoot)(Registered Trademark)rinyah Health Centers
Sampling Method: Non-Probability Sample
Enrollment: 3392 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Estimate of the seasonal burden of Plasmodium falciparum infection among pregnant women and otherwise healthy infants | 3 years
  seasonal burden of Plasmodium falciparum infection

SECONDARY OUTCOMES:
Estimate of the frequency of parasitemia due to non-falciparum malaria | 3 years
  The frequency of parasitemia due to non-falciparum malaria and seroprevalence of parasitic infections due to organisms other than Plasmodium (e.g. filarial spp., Schistosoma spp., soil-transmitted helminths) in these cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Patrick E Duffy, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Maferinyah Rural Health Training and Research Center, Maferinyah, Guinea

REFERENCES:
- [Background] Kwan JL, Seitz AE, Fried M, Lee KL, Metenou S, Morrison R, Kabyemela E, Nutman TB, Prevots DR, Duffy PE. Seroepidemiology of helminths and the association with severe malaria among infants and young children in Tanzania. PLoS Negl Trop Dis. 2018 Mar 26;12(3):e0006345. doi: 10.1371/journal.pntd.0006345. eCollection 2018 Mar. PMID 29579050
- [Background] Rogerson SJ, Desai M, Mayor A, Sicuri E, Taylor SM, van Eijk AM. Burden, pathology, and costs of malaria in pregnancy: new developments for an old problem. Lancet Infect Dis. 2018 Apr;18(4):e107-e118. doi: 10.1016/S1473-3099(18)30066-5. Epub 2018 Jan 31. PMID 29396010